CLINICAL TRIAL: NCT05974254
Title: Auricular Acupuncture As Part Of A Multimodal Regimen For Reduction Of Opioid Analgesic Use After Distal Radius Open Reduction and Internal Fixation- A Randomized Controlled Trial
Brief Title: Auricular Acupuncture As Part Of A Multimodal Regimen After Distal Radius Open Reduction and Internal Fixation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Jaime Ortiz, Professor of Anesthesiology, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-53875
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Radius Fracture Distal; Pain, Postoperative
MeSH Terms: conditions — Wrist Fractures; Pain, Postoperative | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial Group 1 - acupuncture treatment Group 2 - no acupuncture treatment 70 patients per group
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients will be under sedation in the operating room and will not be aware of which treatment group they are in.
  The PACU team and outcomes assessor will not be aware of patient group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Electroauricular acupuncture (Experimental): Immediately after Level 2 sedation is achieved, an enhanced auricular trauma protocol (ATP) will be administered on the ear ipsilateral to the operative side at 8 ear points (Hypothalamus, Amygdala, Hippocampus, Prefrontal Cortex, Point Zero, Shen Men, Insula, Vagus) as described by Cheng (2022). The original ATP was described by Helms (2011). Seirin L 0.2 x 30 mm needles will be placed at Hypothalamus and Shen Men points. Seirin J 0.18 x 15 mm needles will be placed at Amygdala, Hippocampus, Prefrontal Cortex, Point Zero, Vagus, and Insula points. Electrostimulation using an ITO ES 130 microstimulator at 30 HZ with Level 4 intensity, will be applied with the positive lead (red) on Hypothalamus and negative lead (black) at Shen Men for 60 minutes. All needles will be removed 1 hour after insertion.
  Interventions: Device: Acupuncture
- No acupuncture (No Intervention): No acupuncture treatment given

INTERVENTIONS:
Device: Acupuncture — Electroacupuncture
  Arms: Electroauricular acupuncture

SUMMARY:
This randomized controlled trial will test the hypothesis that patients receiving an intraoperative auricular acupuncture protocol will require less postoperative opioid analgesic use compared to those who do not receive acupuncture in the setting of a multimodal analgesic protocol for patients receiving surgery to repair distal radius fractures at a Level 1 trauma center under brachial plexus anesthesia with sedation.

ELIGIBILITY:
Inclusion Criteria:

* Patient ages 18-64
* American Society of Anesthesiologists Physical Status 1, 2, or 3
* Patients scheduled to undergo distal radius ORIF under brachial plexus nerve block

Exclusion Criteria:

* Renal dysfunction (Serum Cr > 1.2) - excluded due to potential for altered metabolism of anesthetic and perioperative medications
* Allergy to any of the standard anesthetic agents
* Patient inability to properly communicate with investigators
* Patient or surgeon refusal

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Total opioid analgesic use for 14 days after surgery | 14 days
  Total opioid given in hospital and taken at home, converted to oral morphine equivalents

SECONDARY OUTCOMES:
Pain scores | 14 days
  Pain scores in PACU and at the 7 and 14 day mark post surgery
Incidence of side effects associated with opioid use | 14 days
  PONV, pruritus, headache, constipation, urinary retention, fatigue, difficulty with concentration, drowsiness, lightheadedness, dry mouth

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Ortiz, MD, MBA, Principal Investigator — Baylor College of Medicine
Locations (1):
- Ben Taub Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No